CLINICAL TRIAL: NCT04699734
Title: Peripheral Nerve Block in Patients With Painful Diabetic Polyneuropathy: How Important is the Peripheral Signaling?
Brief Title: Peripheral Nerve Block in Patients With Painful Diabetic Polyneuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: BPN2020
Record Dates: First submitted 2021-01-04; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Painful Diabetic Neuropathy; Neuropathic Pain; Neuropathy;Peripheral
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia; Neuritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xylocaine (Active Comparator): Nerve block
  Interventions: Diagnostic Test: Xylocaine 1%
- Isotonic saline (Placebo Comparator): Nerve block
  Interventions: Diagnostic Test: NaCl 9mg/ml

INTERVENTIONS:
Diagnostic Test: Xylocaine 1% — Nerve block
  Arms: Xylocaine
Diagnostic Test: NaCl 9mg/ml — Nerve block
  Arms: Isotonic saline

SUMMARY:
The purpose of the present study is to evaluate the role of peripheral afferent input for spontaneous pain in painful diabetic polyneuropathy

DETAILED DESCRIPTION:
Both peripheral and central changes in the nervous system contribute to the development of painful diabetic neuropathy, but how these changes contribute to the pain generation remains yet to be fully understood.

The purpose of this study is to evaluate if a peripheral regional nerve block relieves spontaneous pain in painful diabetic polyneuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Probably diabetic neuropathy confirmed using the Toronto criteria in a "conservative manner", i.e. three out of three symptoms/signs of neuropathy must be present (sensory neuropathy symptoms, distal reduced sensibility, reduced ankle reflexes) 7.
* Definite or probable neuropathic pain for minimum the last 6 months
* Mean pain intensity at > 4 NRS the last week17.

Since we expect a large effect of the block it is not necessary to discontinue pain medication.

Exclusion Criteria:

* Other causes of pain in the same area or other pain that cannot be distinguished from the neuropathic pain.
* Unable to understand and speak Danish.
* Non-cooperative.
* Warfarin or other medication that contraindicate regional anesthesia.
* Infection in the injection area.
* Allergy to lidocaine.
* Pregnancy or lactating (fertile women must to show negative pregnancy test or use anticonception).
* Severe psychiatric disease e.g. severe depression during the last 6 months.
* Alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Indication of pain relieved extremity | 30 minutes
  Number of participants who indicated the leg with lidocaine as most pain relieved 30 minutes after block And number of participants who indicated the leg with saline as most pain relieved 30 minutes after block

SECONDARY OUTCOMES:
Pain intensity | 90 minutes
  Intensity of spontaneous pain (Numeric Rating Scale (NRS) 0-10, 0=no pain 10=worst pain imaginable) 30, 45, 60 and 90 minutes after block
Hyperalgesia and allodynia | 90 minutes
  Intensity of hyperalgesia and allodynia from -5 to 5 (-5 = no sensation, 0=normal sensation, 5=extremely intense sensation) to brush, pinprick, cold and warm at baseline and if there is registered any signs of hyperexcitability at baseline then 35, 60 and 90 minutes after nerve block.
Pain relief | 45 minutes
  Pain relief at 45 minutes after block assessed using a 6-point scale compared to pain intensity at baseline. (-1 = worse pain 0=no relief 1= little 2= moderate 3=good 4=complete)
Pain symptomps | 50 minutes
  Intensity of neuropathic pain symptoms 50 minutes after nerve block Burning: NRS (0-10), 0=no burning 10=worst burning imaginable Squeezing: NRS (0-10), 0=no squeezing 10=worst squeezing imaginable Pressure: NRS (0-10), 0=no pressure 10=worst pressure imaginable Tingling: NRS (0-10), 0=no tingling 10=worst tingling imaginable
Distribution of evoked pain | 60 minutes
  The distribution of any evoked pain to brush, pinprick, cold and warm before and 60 minutes after nerve block will be mapped using a filt pen and afterwards photographed.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen L Schaldemose, MD, Principal Investigator — Danish Pain Research Center, Aarhus University
Locations (1):
- Danish Pain Research Center, Aarhus University, Aarhus University Hospital, Aarhus N, Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tesfaye S, Boulton AJ, Dyck PJ, Freeman R, Horowitz M, Kempler P, Lauria G, Malik RA, Spallone V, Vinik A, Bernardi L, Valensi P; Toronto Diabetic Neuropathy Expert Group. Diabetic neuropathies: update on definitions, diagnostic criteria, estimation of severity, and treatments. Diabetes Care. 2010 Oct;33(10):2285-93. doi: 10.2337/dc10-1303. PMID 20876709